CLINICAL TRIAL: NCT03563118
Title: Evaluation of Prolidase as an Oxidative Stress Marker in Obstructive Sleep Apnea Syndrome
Brief Title: Evaluation of Prolidase in Obstructive Sleep Apnea Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva Sayhan, assiatant prof., Sakarya University
Other Study IDs: OSAS
Record Dates: First submitted 2018-06-07; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep-Apnea Syndrome
Keywords: Prolidase Activity; Obstructive Sleep-Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group OSAS: We included 56 with OSAS [13 subjects 23.2% mild, 19 subjects 33.9% moderate, 24 subjects 42.8% severe
- control group: simple snoring

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent breathing disorder in sleep. We have aimed to evaluate the relationship between OSA and prolidase activity, the oxidative stress index (OSI), total antioxidative capacity (TAC), and total oxidative capacity (TOC) and the relationship between carotid intima media thickness (CIMT).

DETAILED DESCRIPTION:
This study was approved by the local ethics committee in accordance with the Helsinki Declaration. Written informed consent was received from the OSAS Subjects patients and control subjects before enrolment in the study. The patient and control cohorts were recruited from the Pulmonary Medicine Department, Medical Faculty, Yuzuncu Yıl University. Blood samples were analysed at the Biochemistry Laboratory of Harran University Medical Faculty TAC and TOS levels were measured by using an automated measurement method. TAC measurement method involves the production of a potent biological hydroxyl radical. Ferrous ion solution is mixed with hydrogen peroxide. Thus, it is possible to measure the anti-oxidative effect of the sample against the potent free radical reactions initiated by the production of the hydroxyl radical. TOS method is based on the oxidation of ferrous ion to ferric ion in the presence of various oxidant species in acidic medium and the measurement of the ferric ion by xylenol orange. mmol Trolox equivalent (equiv)/L, mmol H2O2 /L and mg/dL, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with OSA after night polysomnography (PSG).
* Patients were enrolled in the study following receipt of their written informed consent.

Exclusion Criteria:

* Patients had ischaemic cardiovascular diseases,
* Patients had chronic obstructive pulmonary diseases,
* Patients had ischaemic cerebral diseases,
* Patients had chronic inflammatory diseases,
* Patients had chronic and acute systemic infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient (male/female: 43/31) were diagnosed with OSA after night polysomnography (PSG)
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Prolidase activity | 1 month
  Prolidase activity was determined by a photometric method based on the measurement of the proline levels produced by prolidase (26). Plasma samples (100ml) were blended with 100 ml of serum physiological. A total of 25 ml of the mixture was preincubated with 75ml of the preincubation solution (50 mmol/l Tris HCl buffer pH 7.0 containing 1mmol/l glutathion, 50mmol/l MnCl2) at 37˚C for 30min.

CONTACTS AND LOCATIONS:
Overall Officials: Havva Sayhan, Study Chair — Sakarya University Research and Training Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Sakarya University Research and Training Hospital, Sakarya, Merkez
  - Sakarya University Research and Training Hospital, Sakarya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yamauchi M, Nakano H, Maekawa J, Okamoto Y, Ohnishi Y, Suzuki T, Kimura H. Oxidative stress in obstructive sleep apnea. Chest. 2005 May;127(5):1674-9. doi: 10.1378/chest.127.5.1674. PMID 15888845